CLINICAL TRIAL: NCT03621852
Title: Prospective Evaluation of the Diagnostic Efficacy of a EUS Guided FNB Needle (AQUIRE®) in Tumors of the Pancreas, Submucosal Tumors and Lymph Node Disease of the Upper GI Tract
Brief Title: Prospective Evaluation of the Diagnostic Efficacy of a EUS Guided FNB Needle (AQUIRE®)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Ulrike Denzer, Prof. Dr. med. Ulrike Denzer, Head of the department of endoscopy, Philipps University Marburg
Other Study IDs: VERSION 2 04/2017
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Tumors of the Pancreas; Submucosal Tumor of Gastrointestinal Tract (Disorder); Lymph Node Disease
Keywords: Endosonography; fine needle biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Endoultrasound guided FNB: Patients with tumors of the pancreas, submucosal tumors or lymphnode disease of the upper gastrointestinal tract, which have to undergo EUS guided FNB.
  Interventions: Device: Endoultrasound guided FNB

INTERVENTIONS:
Device: Endoultrasound guided FNB — EUS FNB with Aquire TM device
  Other Names: EUS FNB with Aquire TM device

SUMMARY:
The present study investigates the efficacy of a new Endoultrasound guided fine needle biopsy (EUS-FNB) device (AquireTM Boston Scientific= AQUIRE®) for obtaining histological tissue cylinders in the diagnosis of solid pancreatic tumors, submucosal tumors of the upper gastrointestinal tract (esophagus, stomach, duodenum) and lymph node disease..

DETAILED DESCRIPTION:
The AquireTM FNB device uses a triple point tip that is designed to maximize tissue capture and minimize fragmentation.

The efficiency of the 22 Gauge needle is evaluated in a prospective single arm study. The material obtained will be collected for formalin fixation and analyzed by a pathologist blinded for the type of needle device.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Indication for EUS FNB with solid pancreatic tumors, submucosal tumors or lymph node disease of the upper gastrointestinal tract will be included

Exclusion Criteria:

* Cystic pancreatic tumors
* Contraindication for EUS FNB
* Lesion of interest cannot be reached endosonographically

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing EUS FNB with solid pancreatic tumors, submucosal tumors or lymph node disease of the upper gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
tissue yield | 12 month after FNB
  The primary outcome of the present study is to analyze the percentage in which a representative histological sample can be obtained by EUS-FNB (quality score 3 as defined by Payne et al.).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätskliniken Gießen und Marburg, Standort Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No